CLINICAL TRIAL: NCT03991715
Title: Sustaining Physical Activity Following Cardiac Rehabilitation Completion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-3306; UL1TR001111 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Rehabilitation
MeSH Terms: interventions — Fitness Trackers

STUDY DESIGN:
Intervention Model Description: This is a pilot study. All participants receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Activity Tracker (Experimental): Participants provided an activity tracker to wear and weekly reports
  Interventions: Behavioral: Activity Tracker

INTERVENTIONS:
Behavioral: Activity Tracker — Individually tailored daily and weekly physical activity goals established for all participants. Participants sent weekly reports for 6 weeks after cardiac rehabilitation discharge.
  Other Names: Fitbit

SUMMARY:
Cardiac rehabilitation participants will be enrolled during cardiac rehabilitation and provided an activity tracker to use.

DETAILED DESCRIPTION:
Cardiac rehabilitation participants will be enrolled during cardiac rehabilitation and provided an activity tracker to use. Each week they will be provided a summary report of their steps and physical activity, that will continue to 6 weeks post discharge from cardiac rehabilitation.

ELIGIBILITY:
Inclusion criteria:

* coronary heart disease
* currently attending cardiac rehabilitation with at least 4 weeks left
* >=18 years of age
* own a smart phone and able to participate in mobile health program
* able to understand and write English
* adequate clinical stability
* understand and sign informed consent

Exclusion criteria:

* currently using a digital physical activity tracker
* past use of a digital activity tracker
* planning to relocate in 12 weeks
* acute coronary artery disease symptoms
* decompensated heart failure
* New York Heart Association class IV heart failure
* severe valvular heart disease
* severe pulmonary hypertension
* cardiac transplantation
* visually impaired, severe
* end stage renal disease
* impairment from stroke, injury, or other medical disorder that precludes participation
* dementia that precludes ability to participate and follow protocol
* inability or unwillingness to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Evenson, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Time Frame: Deidentified individual data that supports the activity tracker results may be shared from 0-12 months following publication.
  Access Criteria: An investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Activity Tracker
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Activity Tracker
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 61.8 [51 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Average Steps Per Day (Preintervention Period)
Description: Average steps per day measured by the activity tracker
Time Frame: pre-intervention (during cardiac rehab starting on the day the tracker was given to cardiac rehab discharge), a total of up to 10 weeks
Population: One participant did not return to cardiac rehabilitation after the enrollment visit (after receiving activity tracker).
Measure: Mean (Full Range); unit: steps per day
Arm/Group | Activity Tracker
Number analyzed (Participants) | 4
steps per day | 6507 [3523 to 9052]

2. Primary Outcome: Average Physical Activity in Minutes Per Day (Preintervention Period)
Description: Average "very active" minutes per day of physical activity measured by the activity tracker
Time Frame: as for outcome 1
Population: One participant did not return to cardiac rehabilitation after the enrollment visit (after receiving activity tracker).
Measure: Mean (Full Range); unit: minutes per day
Arm/Group | Activity Tracker
Number analyzed (Participants) | 4
minutes per day | 14 [2 to 34]

3. Primary Outcome: Average Steps Per Day (Intervention Period)
Description: Average steps per day measured by the activity tracker
Time Frame: Intervention (day following cardiac rehab discharge to the day the last weekly report was sent), a total of up to 10 weeks
Population: One participant did not return to cardiac rehabilitation after the enrollment visit (after receiving activity tracker).
Measure: Mean (Full Range); unit: steps per day
Arm/Group | Activity Tracker
Number analyzed (Participants) | 4
steps per day | 5960 [2828 to 8645]

4. Primary Outcome: Average Physical Activity in Minutes Per Day (Intervention Period)
Description: Average "very active" minutes per day of physical activity measured by the activity tracker
Time Frame: as for outcome 3
Population: One participant did not return to cardiac rehabilitation after the enrollment visit (after receiving activity tracker).
Measure: Mean (Full Range); unit: minutes per day
Arm/Group | Activity Tracker
Number analyzed (Participants) | 4
minutes per day | 11 [2 to 26]

5. Primary Outcome: Average Steps Per Day (Maintenance Period)
Description: Average steps per day measured by the activity tracker
Time Frame: Maintenance (day following when the last weekly report was sent to last day of tracking by staff), a total of up to 15 weeks
Population: One participant did not return to cardiac rehabilitation after the enrollment visit (after receiving activity tracker).
Measure: Mean (Full Range); unit: steps per day
Arm/Group | Activity Tracker
Number analyzed (Participants) | 4
steps per day | 5158 [2819 to 8852]

6. Primary Outcome: Average Physical Activity Per Day (Maintenance Period)
Description: Average "very active" minutes per day of physical activity measured by the activity tracker
Time Frame: Maintenance (day following when the last weekly report was sent to last day of tracking by staff), an overall total of up to 15 weeks
Population: One participant did not return to cardiac rehabilitation after the enrollment visit (after receiving activity tracker).
Measure: Mean (Full Range); unit: minutes per day
Arm/Group | Activity Tracker
Number analyzed (Participants) | 4
minutes per day | 7 [1 to 20]

ADVERSE EVENTS:
Time Frame: From the time of enrollment (approximately 4 weeks prior to cardiac rehabilitation discharge) through 6 weeks post cardiac rehabilitation discharge.
Arm/Group | Activity Tracker
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03991715/Prot_SAP_000.pdf